CLINICAL TRIAL: NCT06420557
Title: Unconscious Reduction of Fear Through Decoded Neuro-Reinforcement
Acronym: DecNef
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michelle Craske, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-001604; R33MH135002 (NIH)
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Phobia
Keywords: unconscious fear extinction; anxiety disorders; decoded neuro-reinforcement
MeSH Terms: conditions — Phobic Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 Session (Experimental): 1 neuro-reinforcement session
  Interventions: Behavioral: Unconscious Neuro-reinforcement
- 3 Sessions (Experimental): 3 neuro-reinforcement sessions
  Interventions: Behavioral: Unconscious Neuro-reinforcement
- 5 sessions (Experimental): 5 neuro-reinforcement sessions
  Interventions: Behavioral: Unconscious Neuro-reinforcement

INTERVENTIONS:
Behavioral: Unconscious Neuro-reinforcement — Individuals will complete an implicit fmri neuro-reinforcement task where real-time brain activity is matched to a desired activation. Individuals will also receive financial reward for activating the desired activation. Visual feedback will be presented to indicate how well individuals' brain activity matches the desired activation. Individuals will complete 1 session of neuro-reinforcement.
  Arms: 1 Session
Behavioral: Unconscious Neuro-reinforcement — Individuals will complete an implicit fmri neuro-reinforcement task where real-time brain activity is matched to a desired activation. Individuals will also receive financial reward for activating the desired activation. Visual feedback will be presented to indicate how well individuals' brain activity matches the desired activation. Individuals will complete 3 sessions of neuro-reinforcement.
  Arms: 3 Sessions
Behavioral: Unconscious Neuro-reinforcement — Individuals will complete an implicit fmri neuro-reinforcement task where real-time brain activity is matched to a desired activation. Individuals will also receive financial reward for activating the desired activation. Visual feedback will be presented to indicate how well individuals' brain activity matches the desired activation. Individuals will complete 5 sessions of neuro-reinforcement.
  Arms: 5 sessions

SUMMARY:
This application investigates the efficacy of a novel method of neuro-reinforcement based on decoded fMRI activity to reduce fear responses in individuals with phobias (e.g., spiders, snakes). This method works unconsciously in the brain, without the need for participants to endure repeated conscious exposures to their feared stimuli. Fear-related disorders such as specific phobia, post-traumatic stress disorder (PTSD), and other anxiety disorders present a major challenge, as effective treatment options usually involve repeated exposures to feared stimuli, leading to high levels of distress, fear, and panic that can motivate premature treatment termination. Consequently, there is an unmet need for treatment that minimizes subjective discomfort and attrition in order to maximize efficacy. Recent developments in computational neuroimaging have enabled a method that can deliver unconscious exposure to feared stimuli, resulting in effective fear reduction while bypassing a primary cause of treatment attrition. Because this treatment method happens unconsciously in the brain, changes in behavior outcomes are potentially more likely to generalize to different contexts, thereby overcoming a limitation of traditional treatments.

DETAILED DESCRIPTION:
The gold standard treatment for specific phobias is exposure therapy, wherein the individual repeatedly faces the object of their fear. However, for many patients, the level of distress prohibits them from either starting or completing exposure therapy. The objective of this application is to use focal neuro-reinforcement based on decoded fMRI information (from the ventral temporal temporal cortex) to reduce fear responses to feared animal stimuli (e.g., spiders, birds) in individuals with phobias, directly and unconsciously in the brain, without repeatedly consciously exposing participants to their feared stimuli. Because the induced representations are unconscious, participants do not experience negative emotional responses and the procedure is double-blind placebo-controlled, thus providing a level of experimental rigor not afforded to standard psychological therapies. Extending from our pilot data, we are positioned to test the mechanisms and behavioral outcomes of a novel treatment for phobias that at the same time advances our understanding of the role of consciousness in fear responses and their change over time. The specific aims are to: (1) confirm that our method engages the neurobiological target (amygdala reactivity to images of feared animals) in a population of individuals with specific phobias of animals; (2) quantify how changes in amygdala reactivity with neuro-reinforcement mediate changes in behavioral outcomes, as measured by attentional capture, approach/avoidance behavior, or subjective fear ratings, immediately post neuro-reinforcement; (3) assess the longer term effects four weeks after neuro-reinforcement; and (4) explore the impact of three dosage levels of neuro-reinforcement to identify the optimal dosage for future research. If proven effective, the results will inform applications for other fear related disorders, such as posttraumatic stress disorder, social anxiety disorder and panic disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Individual has normal or corrected to normal vision
2. Individual has normal or corrected to normal hearing
3. Individual is competent to understand informed consent
4. Individual must meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for specific phobias, animal subtype

Exclusion Criteria:

1. Individual is unable to fill in consent form correctly
2. Individual is unable to respond adequately to screening questions
3. Individual is unable to maintain focus or to sit during assessment
4. Individual has history of: neurological disease or defect (e.g., stroke, traumatic brain injury, schizophrenia or other psychological disorders, or seizures) Individual has vision problems (including cataracts, amblyopia, or glaucoma) Individual presents with: Obsessive Compulsive Disorder, Substance Use Disorder, Bipolar Disorder, Psychosis, neurologic diagnoses or unstable serious medical conditions
5. Participant receives an elevated score on the PHQ-9
6. Individual does not present with more than one object of specific phobia
7. Individual can touch the phobic object category during the pre-treatment Behavioral Approach Test without presenting significant distress
8. Individual is currently prescribed psychotropic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Amygdala Reactivity | 14 days (measured at pre-treatment and 2 weeks)
  The neural measure of difference in amygdala reactivity (measured by fMRI) to target phobic animals compared to control phobic animals from pre-treatment to post-treatment. Lower numbers (i.e. more negative numbers) indicate greater amygdala decrease and and better outcomes.
Subjective Fear Post-treatment Minus Pre-treatment | 14 days (measured at pre-treatment and 2 weeks)
  Subjective Fear Ratings of images of targeted phobic stimuli Minimum score of 0, Maximum score of 180, higher scores mean worse outcome.

SECONDARY OUTCOMES:
Skin Conductance Response: Physiological Arousal Post-treatment Minus Pre-treatment | 14 days (measured at pre-treatment and 2 weeks)
  Skin conductance to image presentation of targeted phobic stimuli post-treatment minus pre-treatment
Fear Survey Schedule | 14 days (measured at pre-treatment and 2 weeks)
  Subjective fear ratings of a list of typical phobic stimuli Minimum score of 40, maximum of 200, higher scores mean worse outcome.
Stroop Task Post-treatment Minus Pre-treatment | 14 days (measured at pre-treatment and 2 weeks)
  Measure of preferential allocation of attentional resources measured in reaction time (seconds) for visual presentation of the targeted phobic stimulus
Approach/Avoidance Behavior in VR Post-treatment Minus Pre-treatment | 14 days (measured at pre-treatment and 2 weeks)
  Maximal approach distance will be assessed in a behavioral approach test conducted in a virtual reality context. The Behavioral Approach Test follows a ten-step procedure of increasing difficulty to approach a feared animal (e.g. snakes), beginning with a first step such as standing in the same room as the feared animal. Then, participants approach the feared animal step-by-step, taking time at each step, until a final step such as holding the feared animal or having it touch you is reached. Behavioral outcomes that will be measured from the Behavioral Approach Test include a) maximal approach distance and b) subjective fear ratings at each distance. Minimum score for approach distance is 1, and highest is 10 (numbers represent steps taken toward fearful stimulus). Higher scores represent a better outcome on this task.
Subjective Fear Ratings in Virtual Reality (VR) Post-treatment Minus Pre-treatment | 14 days (measured at pre-treatment and 2 weeks)
  Subjective fear ratings will be assessed at each distance in a behavioral approach test conducted in a virtual reality context. The Behavioral Approach Test follows a ten-step procedure of increasing difficulty to approach a feared animal (e.g. snakes), beginning with a first step such as standing in the same room as the feared animal. Then, participants approach the feared animal step-by-step, taking time at each step, until a final step such as holding the feared animal or having it touch you is reached. Minimum score for subjective fear is 1, and maximum is 8. Higher scores represent a worse outcome on this task.
Patient Health Questionnaire (PHQ-9) | 14 days (measured at pre-treatment and 2 weeks)
  Self-reported depression severity. Scores range from 0-27, with higher scores indicating greater severity.
Generalized Anxiety Disorder-7 (GAD-7) | 14 days (measured at pre-treatment and 2 weeks)
  Self-reported anxiety severity. Scores range from 0-21, with higher scores indicating greater severity.
Severity of Phobias questionnaire | 14 days/6 weeks (measured at pre-treatment, 2 weeks, and 6 weeks)
  Self-report severity of phobias rating; 10 items. Scores range from "Never" to "All of the time," with a higher score indicating greater severity.
Behavioral Inhibition/Behavioral Activation Scales (BIS/BAS) | 0 days (measured at pre-treatment)
  Self-report behavioral inhibition/activation rating; 20 items. Scores range from "Very true for me" to "Very false for me," with a higher score indicating greater severity.
Vividness of Visual Imagery Questionnaire (VVIQ) | 0 days (measured at pre-treatment)
  Self-report vividness of visual imagery; 16 items. Scores range from "No image at all, you only "know" that you are thinking of the object" to "Perfectly real and vivid as real seeing," where higher scores indicate greater vividness of imagery.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G Craske, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States